CLINICAL TRIAL: NCT04954131
Title: A Multi-center, Double-blind, Randomized, Controlled, Phase 2 Study to Evaluate the Immunogenicity and Safety of CpG 1018/Alum-adjuvanted Recombinant SARS-CoV-2 Trimeric S-protein Subunit Vaccine (SCB-2019) in Individuals Aged 18 Years and Older in China
Brief Title: Immunogenicity and Safety Study of Adjuvanted SARS-CoV-2 (SCB-2019) Vaccine in Adultsin China
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhejiang Clover Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CLO-SCB-2019-010
Record Dates: First submitted 2021-07-06; First posted 2021-07-08 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — SCB-2019 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCB-2019 vaccine (Experimental): Investigational SCB-2019 vaccine contains 30 μg of SCB-2019 antigen, and 1.5 mg CpG 1018 and 0.75 mg Alhydrogel as adjuvants, in each 0.5 mL dose
  Interventions: Biological: Candidate Vaccine, SCB-2019
- Placebo (Placebo Comparator): Saline solution (0.9%)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Candidate Vaccine, SCB-2019 — 30 μg of SCB-2019 antigen, and 1.5 mg CpG 1018 and 0.75 mg Alhydrogel as adjuvants
  Arms: SCB-2019 vaccine
Other: Placebo — Saline solution (0.9%)
  Arms: Placebo

SUMMARY:
The purpose of this clinical study, CLO-SCB-2019-010, is to assess the immunogenicity, reactogenicity and safety of the SCB-2019 vaccine in Chinese participants, and to show the comparability of the immune response versus randomly selected individuals who participated in the large-scale efficacy study with the SCB-2019 vaccine (Study CLO-SCB-2019-003).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age.
2. Individuals are willing and able to comply with study requirements, including all scheduled visits, vaccinations, laboratory tests and other study procedures.
3. Individuals are willing and able to give an informed consent, prior to screening.
4. Healthy participants or participants with pre-existing medical conditions who are in a stable medical condition. (A stable medical condition is defined as medication not requiring major change for specific past medical condition, not receive surgery or minimal invasive medical intervention, and without hospitalization or ER visit during the 3 months before enrollment.)
5. Female participants of childbearing potential may be enrolled in the study, if the participant has practiced adequate contraception for 30 days prior to vaccination, and has a negative pregnancy test on the day of vaccination and has agreed to continue adequate contraception for 6 months after the last vaccination.
6. Male participants must agree to employ acceptable contraception from the day of the first dose of the study vaccine/placebo until 6 months after the last dose of the study vaccine/placebo and also refrain from donating sperm during this period.

Exclusion Criteria:

1. Individuals with fever >37.3°C (axillary), or any acute illness at baseline (Day 1) or within 3 days prior to randomization. Participants meeting this criterion may be rescheduled within the relevant window. Febrile participants with minor illnesses can be enrolled at the discretion of the investigator.
2. Individuals with laboratory-confirmed SARS-CoV-2 infection [as defined by reverse transcriptase polymerase chain reaction (RT-PCR) assay or Rapid COVID-19 Antigen Test or an equivalent at Visit 1] or with history of COVID-19, or individual with COVID-19 pandemic area contaction confirmed with inspection or health code on cellphone.
3. Individuals who have received an investigational or authorized COVID-19 vaccine prior to Day 1, or plan to receive COVID-19 vaccine during the study period.
4. Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease [e.g., malignancy, human immunodeficiency virus (HIV) infection] or immunosuppressive/cytotoxic therapy (e.g., systemic corticosteroids, medications used for cancer chemotherapy, organ transplantation or to treat autoimmune disorders) within 3 months prior to Day 1.
5. Individuals with any progressive unstable or uncontrolled clinical conditions.
6. Individuals who are pregnant, or breastfeeding, or planning to become pregnant while enrolled in this study or during the study period.
7. Individuals who have a history of severe adverse reaction associated with a vaccine or severe allergic reaction [e.g., anaphylaxis to any component of the study vaccines (CpG 1018, aluminum), or SCB-2019 components as outlined in the latest IB].
8. Individuals who have a history of malignancy within 1 year before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix which have been cured, or other malignancies with minimal risk of recurrence).
9. Individuals who have received any other investigational product within 30 days prior to Day 1 or intend to participate in another clinical study at any time during the conduct of this study.
10. Individuals who have received any other licensed vaccines within 14 days prior to enrollment in this study or who are planning to receive any vaccine up to Day 53.
11. Individuals with known bleeding disorder that would, in the opinion of the investigator, contraindicate intramuscular injection.
12. Individuals who have received treatment with Rituximab or any other anti-CD20 monoclonal antibodies within 9 months prior to Day 1 or planned during the study period.
13. Administration of intravenous immunoglobulins and/or any blood products within 3 months prior to enrollment or planned administration during the study period.
14. Individuals with any condition that, in the opinion of the investigator, would interfere with the primary study objectives or pose additional risk to the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 766 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
GMT ratio of GMT-CLO-SCB-2019-010 over GMT-CLO-SCB-2019-003 | Day 36
  To demonstrate that SCB-2019 vaccine in this study of Chinese participants elicits immune response that is non-inferior to that in a randomly selected subset of participants of the CLO-SCB-2019-003 clinical study, as measured by virus neutralization assay

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanxi Center for Disease Control and prevention, Taiyuan, Shanxi
  - Sichuan Center for disease control, Chengdu, Sichuan